CLINICAL TRIAL: NCT03516227
Title: Effects of Biofeedback Combined With Abdominal Breathing on Physiological and Psychological Aspects in Patients With Acute Cerebral Infarction
Brief Title: Effects of Biofeedback in Patients With Acute Cerebral Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Yu-Ju Chen, Assistant Professor, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NDMCTaiwan
Record Dates: First submitted 2018-04-23; First posted 2018-05-04 (Actual); Results first posted 2019-10-11 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-09

CONDITIONS: Acute Ischemic Stroke; Biofeedback; Autonomic Dysfunction, Cognitive Function; Psychological Distress
MeSH Terms: conditions — Ischemic Stroke; Primary Dysautonomias

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRVBF (Experimental): Heart rate variability biofeedback
  Interventions: Behavioral: heart rate variability biofeedback
- Control (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: heart rate variability biofeedback — The HRVBF group received four, one-on-one bedside biofeedback training sessions (20-minutes a day for 4 days), and practiced on their own (10-minutes twice a day) using a FDA-regulated, hand-held mobile biofeedback device (StressEraser, Helico Inc., New York, NY, USA).26 The control group received usual care.Afterwards, all participants were telephoned bi-weekly and encouraged to practice slow breathing (HRVBF group) or to perform self-care (control group) for three months.
  Arms: HRVBF

SUMMARY:
The major aim of this study is to investigate the effects of biofeedback assisted abdominal breathing training on improving the psychological and physiological distress in patients with ACI. In this randomized, controlled, single-blind trial, AIS patients were randomly assigned into experimental and control groups. The experimental group received four HRVBF training sessions. The control group received routine care. Repeated measures of HRV, Mini-Mental Status Examination (MMSE), Hospital Anxiety and Depression Scales (HADS), and Barthel Index for ADLs were collected prior to, and at one, and three months post-intervention.

DETAILED DESCRIPTION:
Study protocol Participants who provided signed consent were randomly assigned to HRVBF intervention or control group. They underwent baseline measurements of demographics, psychological distress, cognitive impairment, ADL capabilities, and autonomic function. Random numbers from the Bernoulli distribution were calculated using the Excel BINOMDIST function, and concealed in an opaque envelope, until participants' baseline measurements were completed.

The HRVBF group received four, one-on-one bedside biofeedback training sessions (20-minutes a day for 4 days), and practiced on their own (10-minutes twice a day) using a FDA-regulated, hand-held mobile biofeedback device (StressEraser, Helico Inc., New York, NY, USA).26 The control group received usual care. Afterwards, all participants were telephoned bi-weekly and encouraged to practice slow breathing (HRVBF group) or to perform self-care (control group) for three months. psychological distress, cognitive impairment, ADL capabilities, and autonomic function (represented by HRV) were re-assessed at one, and 3-months after the intervention, by an independent investigator blinded to group assignment.

HRVBF intervention protocol The HRVBF protocol was modified from Lehrer's HRV biofeedback manual.20 A noninvasive visual biofeedback system (NeXus-10 with BioTrace+, Mind Media B.V., Netherlands) and a laptop computer were used for the intervention. Participants in the HRVBF group received four, one-on-one bedside training sessions (20-minutes a day for 4 days). The first session (Day 1) was focused on teaching patients to breath slowly (6-8 breaths-per-minute) and to extend their expiratory phase using pursed-lip breathing. Also, respiration sensors for tracking breathing pace were introduced. The second session (day 2) was focused on teaching patients diaphragmatic breathing in conjunction with pursed-lip breathing, and to use respiratory sensors to pace breathing (6 breaths a minute). The third and fourth sessions (days 3 and 4) were focused on reviewing diaphragmatic breathing, pursed-lip breathing, and teaching patients to breathe in-phase with their heart rate changes. Additionally, participants were encouraged to practice slow diaphragmatic and pursed-lip breathing, on their own, with the aid of the hand-held biofeedback device, for 10 minutes, twice-a-day, during the 4-day training period.

ELIGIBILITY:
Inclusion Criteria:

* patients within one week of their first ever ischemic stroke, who were 20 years of age or older, and who were able to express themselves through oral or written communication.

Exclusion Criteria:

* Patients diagnosed with cardiac arrhythmia, mental illness, dementia or Alzheimer's disease, or totally paralyzed and totally dependent on others for care

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-11-09 (Actual); Primary Completion 2016-06-26 (Actual); Study Completion 2016-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Ju Chen, Ph.D., Principal Investigator — National Defense Medical Center

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the neurological ward at a medical center in northern Taiwan.
Pre-assignment Details: Five patients did not receive the allocated group treatment protocol (two had arrhythmias after inclusion and three refused baseline measurements)
Period: Overall Study
Arm/Group | HRVBF | Control
Started | 20 | 20
Completed | 19 | 16
Not Completed | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- HRVBF: Heart rate variability biofeedback
  heart rate variability biofeedback: The HRVBF group received four, one-on-one bedside biofeedback training sessions (20-minutes a day for 4 days), and practiced on their own (10-minutes twice a day) using a FDA-regulated, hand-held mobile biofeedback device (StressEraser, Helico Inc., New York, NY, USA). The control group received usual care.Afterwards, all participants were telephoned bi-weekly and encouraged to practice slow breathing (HRVBF group) or to perform self-care (control group) for three months.
- Total: Total of all reporting groups
Arm/Group | HRVBF | Control | Total
Number analyzed (Participants) | 19 | 16 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (11.4) | 67.2 (7.6) | 67.4 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 10 | 8 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Taiwan | 19 | 16 | 35

OUTCOME MEASURES:

1. Primary Outcome: Changes From Baseline Psychological Distress (Anxiety and Depression) at 1 and 3 Months
Description: The hospital anxiety and depression scale was a 14-item ordinal scale, used for participants to self-rate their psychological distress related to anxiety (7 items) and depression (7 items). Items are scored 0(no distress) to 3 (serious distress). Based on the findings from previous studies, scoring at or higher than the cut-off point of 8 out of 21, identified those with anxiety or depression. The minimum and maximum values of both anxiety and depression are 0 and 21, respectively. The higher scores mean a worse outcome.
Time Frame: baseline, 1-month, and 3-month visits
Population: Thirty-five participants completed all aspects of the study (19 intervention, 16 control)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HRVBF | Control
Number analyzed (Participants) | 19 | 16
score on a scale
  Baseline_Anxiety | 14.74 (4.15) | 14.75 (3.30)
  Baseline_Depression | 13.11 (3.20) | 14.25 (2.97)
  1-month_Anxiety | 12.79 (3.16) | 15.38 (2.09)
  1-month_Depression | 11.53 (4.20) | 15.75 (2.82)
  3-month_Anxiety | 10.58 (2.97) | 12.88 (3.03)
  3-month_Depression | 8.42 (4.99) | 13.25 (4.12)

2. Primary Outcome: Changes From Baseline Cognitive Function at 1 and 3 Months
Description: The Mini-Mental State Examination (MMSE) was used to measure patients' cognitive function. MMSE includes eleven items and consists of five facets orientation (space and time, registration, attention and calculation, recall, and language). The minimum value is 0 and the maximum value is 30. Lower scores represent a worse cognitive function.
Time Frame: baseline, 1-month, and 3-month visits
Population: Thirty-five participants completed all aspects of the study (19 intervention, 16 control)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | HRVBF | Control
Number analyzed (Participants) | 19 | 16
score on a scale
  Baseline_MMSE | 18.84 (3.88) | 20.00 (3.48)
  1-month_MMSE | 21.68 (4.23) | 21.00 (3.46)
  3-month_MMSE | 23.74 (3.86) | 22.38 (3.34)

3. Primary Outcome: Changes From Baseline Capabilities of Activities of Daily Living at 1 and 3 Months
Description: The 10-item Barthel Index (BI) was used to measure participants' capabilities in activities of daily living (ADLs) (feeding, bathing, grooming, dressing, transfers, and toilet use). BI score ranges from 0 to 100 with lower scores indicating lower ADLs capabilities.
Time Frame: baseline, 1-month, and 3-month visits
Population: Thirty-five participants completed all aspects of the study (19 intervention, 16 control)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HRVBF | Control
Number analyzed (Participants) | 19 | 16
score on a scale
  Baseline_BI | 45.00 (24.27) | 45.31 (12.31)
  1-month_BI | 54.47 (23.09) | 54.38 (14.48)
  3-month_BI | 67.11 (22.50) | 65.00 (18.07)

4. Primary Outcome: Changes From Baseline Autonomic Function (Time-domain of Heart Rate Variability) at 1 and 3 Months
Description: Heart rate variability (HRV) was used to represent the autonomic function and measured with Mind Media B.V. (-Nexus-10, Netherlands). Time-domain of HRV was analyzed using Kubios HRV software (Biosignal Analysis and Medical Imaging Group, Finland). Time-domain indices of HRV indices: standard deviation of normal to normal R-R intervals (SDNN) and root mean square of successive heartbeat interval differences (rMSSD), which were reported with the Unit of Measure "ms". The higher scores mean a better outcome.
Time Frame: baseline, 1-month, and 3-month visits
Population: Thirty-five participants completed all aspects of the study (19 intervention, 16 control)
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | HRVBF | Control
Number analyzed (Participants) | 19 | 16
ms
  Baseline_SDNN ln | 2.24 (0.26) | 2.38 (0.18)
  Baseline_rMSSD ln | 2.37 (0.27) | 2.50 (0.15)
  1-month_SDNN ln | 2.44 (0.24) | 2.46 (0.14)
  1-month_rMSSD ln | 2.51 (0.24) | 2.58 (0.17)
  3-month_SDNN ln | 2.47 (0.27) | 2.43 (0.19)
  3-month_rMSSD ln | 2.56 (0.24) | 2.52 (0.19)

5. Primary Outcome: Changes From Baseline Autonomic Function (Frequency-domain of Heart Rate Variability) at 1 and 3 Months
Description: Heart rate variability (HRV) was used to represent the autonomic function and measured with Mind Media B.V. (-Nexus-10, Netherlands). Frequency-domain of HRV was analyzed using Kubios HRV software (Biosignal Analysis and Medical Imaging Group, Finland). Frequency domain indices of HRV were low frequency (LF), high frequency (HF), and total power (TP), which were reported with the unit of Measure "ms^2". The higher scores mean a better outcome.
Time Frame: baseline, 1-month, and 3-month visits
Measure: Mean (Standard Deviation); unit: ms^2
Arm/Group | HRVBF | Control
Number analyzed (Participants) | 19 | 16
ms^2
  Baseline_LF ln | 3.41 (0.87) | 3.79 (0.79)
  Baseline_HF ln | 3.27 (0.55) | 3.51 (0.39)
  Baseline_TP ln | 4.14 (0.63) | 4.44 (0.56)
  1-month_LF ln | 4.08 (0.62) | 3.80 (0.52)
  1-month_HF ln | 3.73 (0.56) | 3.73 (0.47)
  1-month_TP ln | 4.74 (0.56) | 4.58 (0.40)
  3-month_LF ln | 4.01 (0.76) | 3.85 (0.60)
  3-month_HF ln | 3.64 (0.50) | 3.52 (0.51)
  3-month_TP ln | 4.73 (0.58) | 4.59 (0.45)

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Groups:
- HRVBF; Control: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | HRVBF | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No